CLINICAL TRIAL: NCT04051099
Title: Bilateral Superficial Cervical Plexus Block Combined With Intravenous Sedation Versus General Anesthesia in Selected Patients for Thyroid/Parathyroid Surgery ; a Prospective Randomized Control Trial
Brief Title: Bilateral Superficial Cervical Plexus Block in Thyroid/Parathyroid Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Suwimon Tangwiwat, Assistant professor, Department of Anesthesiology, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Si 116/2018
Record Dates: First submitted 2018-03-27; First posted 2019-08-09 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Benign Tumor of Thyroid; Hyperparathyroidism
Keywords: bilateral superficial cervical plexus block; thyroid surgery; parathyroid surgery
MeSH Terms: conditions — Hyperparathyroidism | interventions — Bupivacaine; Dexmedetomidine; Conscious Sedation; Anesthesia, General

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bilateral cervical plexus block (Experimental): bilateral superficial cervical plexus block with 0.25% bupivacaine 8 ml each (total 0.25% bupivacaine 16 mg)
  Interventions: Procedure: Bilateral superficial cervical plexus block with 0.25% bupivacaine 8 ml each (total 16 ml); Drug: Dexmedetomidine plus propofol infusion; Procedure: Local infiltraion analgesia
- General anesthesia (Experimental): General anesthesia with endotracheal intubation under total intravenous anesthesia (TIVA)
  Interventions: Drug: Dexmedetomidine plus propofol infusion; Procedure: Local infiltraion analgesia; Procedure: General anesthesia with endotracheal tube

INTERVENTIONS:
Procedure: Bilateral superficial cervical plexus block with 0.25% bupivacaine 8 ml each (total 16 ml) — bilateral superficial cervical plexus
  Other Names: BSCPB
  Arms: bilateral cervical plexus block
Drug: Dexmedetomidine plus propofol infusion — Dexmedetomidine 0.5 ug/kg infusion in 10 min then 0.5 ug/kg/h, Propofol infusion
  Other Names: Conscious sedation
Procedure: Local infiltraion analgesia — local infiltration analgesia with 2%lidocaine with adrenaline 5 ug/ml 10 ml
  Other Names: LIA
Procedure: General anesthesia with endotracheal tube — Induction with Propofol and intubation with cisatracurium
  Other Names: GA with ETT
  Arms: General anesthesia

SUMMARY:
To compare efficacy and safety between bilateral superficial cervical plexus block combined with intravenous sedation (RA group) and general anesthesia (GA group) for thyroid and parathyroid operations. This study evaluates postoperative numerical pain score and systemic opioid requirement within 24 hours.

DETAILED DESCRIPTION:
According to literature review, there is limit information about efficacy and safety of thyroid and parathyroid operations under bilateral superficial cervical plexus block combined with intravenous sedation without general anesthesia. General anesthesia is commonly used for neck operations because it is easy to perform. However in high cardiovascular or pulmonary risk patients such as end stage renal disease (ESRD) patients, regional anesthesia such as superficial cervical plexus block combined with intravenous sedation have become an alternative technique for neck operations.

This study evaluate whether regional anesthesia (RA) technique can be the alternative technique for thyroid/parathyroid surgery compare to conventional technique (GA).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) grade I-III, aged over 18 years
* Elective thyroidectomy, thyroid lobectomy, parathyroidectomy

Exclusion Criteria:

* Language barrier or inability to communicate with the operating team
* Allergy to local anaesthetic
* Known substernal, retroesophageal or retrotracheal goiter
* Thyroid cancer
* Previous neck exploration or neck radiation
* Recurrent laryngeal nerve paralysis
* BMI ≥ 30

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain score at rest | 0 hour at PACU ( time PACU arrival)
  Numerical rating scale 0-10 (0=no pain, 10= worst pain imaginable)
Postoperative pain score at rest | 1 hours at PACU
  Numerical rating scale 0-10 (0=no pain, 10= worst pain imaginable)
Postoperative pain score at rest | 6 hours at ward
  Numerical rating scale 0-10 (0=no pain, 10= worst pain imaginable)
Postoperative pain score at rest | 12 hours at ward
  Numerical rating scale 0-10 (0=no pain, 10= worst pain imaginable)
Postoperative pain score at rest | 18 hours at ward
  Numerical rating scale 0-10 (0=no pain, 10= worst pain imaginable)
Postoperative pain score at rest | 24 hours at ward
  Numerical rating scale 0-10 (0=no pain, 10= worst pain imaginable)

SECONDARY OUTCOMES:
Postoperative pain score on swallow | 1 hour PACU
  Numerical rating scale 0-10 (0=no pain, 10= worst pain imaginable)
Postoperative pain score on swallow | average NRS at ward at 24 hours
  Numerical rating scale 0-10 (0=no pain, 10= worst pain imaginable)
Postoperative morphine consumption | Cumulative dose within 24 hours
  in milligram
Complications | within 24 hours
  Percentage of patients present with hoarseness, dyspnea, local anaesthetic systemic toxicity
Patient's satisfaction scale score | at 24 hours
  satisfaction scale score 0-10 ( 0= highly unsatisfied, 10= highly satisfied)

OTHER OUTCOMES:
Conversion rate from RA to GA | intraoperation
  Inable operation due to pain or movement, need to convert from RA toGA

CONTACTS AND LOCATIONS:
Overall Officials: Suwimon Tangwiwat, MD, Principal Investigator — Siriraj Hospital
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ueshima H, Hara E, Hiroshi O. RETRACTED: Successful cases of thyroid surgery performed under only bilateral cervical plexus blocks. J Clin Anesth. 2016 Nov;34:206. doi: 10.1016/j.jclinane.2016.04.014. Epub 2016 May 11. No abstract available. PMID 27687375 (Retraction: PMID 35393198 J Clin Anesth. 2022 Aug;79:110731)
- [Background] Wang Q, Li Z, Xu S, Li Y, Zhang X, Liu Q, Xia Y, Papadimos TJ, Xu X. Feasibility of ultrasound-guided capsule-sheath space block combined with anterior cervical cutaneous nerves block for thyroidectomy: an observational pilot study. BMC Anesthesiol. 2015 Jan 19;15(1):4. doi: 10.1186/1471-2253-15-4. eCollection 2015. PMID 25670918
- [Background] Suh YJ, Kim YS, In JH, Joo JD, Jeon YS, Kim HK. Comparison of analgesic efficacy between bilateral superficial and combined (superficial and deep) cervical plexus block administered before thyroid surgery. Eur J Anaesthesiol. 2009 Dec;26(12):1043-7. doi: 10.1097/EJA.0b013e32832d6913. PMID 19571762
- [Background] Cai HD, Lin CZ, Yu CX, Lin XZ. Bilateral superficial cervical plexus block reduces postoperative nausea and vomiting and early postoperative pain after thyroidectomy. J Int Med Res. 2012;40(4):1390-8. doi: 10.1177/147323001204000417. PMID 22971490
- [Background] Ingsathit A, Thakkinstian A, Chaiprasert A, Sangthawan P, Gojaseni P, Kiattisunthorn K, Ongaiyooth L, Vanavanan S, Sirivongs D, Thirakhupt P, Mittal B, Singh AK; Thai-SEEK Group. Prevalence and risk factors of chronic kidney disease in the Thai adult population: Thai SEEK study. Nephrol Dial Transplant. 2010 May;25(5):1567-75. doi: 10.1093/ndt/gfp669. Epub 2009 Dec 27. PMID 20037182
- [Background] Spanknebel K, Chabot JA, DiGiorgi M, Cheung K, Lee S, Allendorf J, Logerfo P. Thyroidectomy using local anesthesia: a report of 1,025 cases over 16 years. J Am Coll Surg. 2005 Sep;201(3):375-85. doi: 10.1016/j.jamcollsurg.2005.04.034. PMID 16125070
- [Background] Yerzingatsian KL. Thyroidectomy under local analgesia: the anatomical basis of cervical blocks. Ann R Coll Surg Engl. 1989 Jul;71(4):207-10. PMID 2774445